CLINICAL TRIAL: NCT05225415
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2, 6-month Study to Evaluate the Safety, Tolerability and Exploratory Efficacy of CT1812 in Subjects With Mild to Moderate Dementia With Lewy Bodies
Brief Title: Study to Evaluate the Safety, Tolerability and Efficacy of CT1812 in Subjects With Mild to Moderate Dementia With Lewy Bodies
Acronym: COG1201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cognition Therapeutics (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COG1201; R01AG071643 (NIH)
Record Dates: First submitted 2022-01-11; First posted 2022-02-04 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Dementia With Lewy Bodies
Keywords: Dementia
MeSH Terms: conditions — Lewy Body Disease; Dementia

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- CT1812 300 mg (Active Comparator): CT1812 300 mg
  Interventions: Drug: CT1812
- CT1812 100 mg (Active Comparator): CT1812 100 mg
  Interventions: Drug: CT1812
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: CT1812

INTERVENTIONS:
Drug: CT1812 — Orally administered CT1812

SUMMARY:
Multi-center, randomized, double-blind, placebo-controlled, 6- month study in subjects with mild to moderate Dementia with Lewy Bodies.

DETAILED DESCRIPTION:
The safety and efficacy of CT1812 at doses of 300 and 100mg will be evaluated over a 24 week double-blind treatment period in patient diagnosed with dementia with Lewy bodies.

Patients will be randomized 1:1:1 to placebo, 100mg CT1812 or 300mg CT1812. Oral CT1812 will be taken daily. Subjects meeting eligibility requirement and signing informed consent will be assessed by repeated psychometric/neurologic testing, safety procedures and PK and PD sample collection at defined intervals throughout the study. Plasma and CSF biomarkers will also be followed.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 50-85 years of age (inclusive), meeting criteria for probable Dementia with Lewy Bodies (DLB).
* MRI, or CT scan due to contraindication of MRI if approved by medical monitor) obtained during screening consistent with the clinical diagnosis of DLB and without findings of significant exclusionary abnormalities. An historical MRI (or CT scan), up to 1 year prior to screening, may be used if there is no history of intervening neurologic disease or clinical events (such as a stroke, head trauma etc.) and the subject is without clinical symptoms or signs suggestive of such intervening events.
* MMSE 18-27 inclusive

Exclusion Criteria:

* Any neurological condition that may be contributing to cognitive impairment above and beyond those caused by the subject's DLB, including any co-morbidities detected by clinical assessment or MRI (or CT scan due to contraindication of MRI, if approved by medical monitor)
* Screening MRI (or historical MRI or CT scan due to contraindication of MRI if approved by medical monitor) or historical MRI/CT scan, if applicable. of the brain indicative of significant abnormality, including, but not limited to, prior hemorrhage or infarct > 1 cm3, >3 lacunar infarcts, cerebral contusion, encephalomalacia, aneurysm, vascular malformation, subdural hematoma, hydrocephalus, space-occupying lesion (e.g. abscess or brain tumor such as meningioma). If a small incidental meningioma is observed, the medical monitor may be contacted to discuss eligibility.
* Clinical, laboratory findings or medical history consistent with:

  1. Other primary degenerative dementia (fronto-temporal dementia, Huntington's disease, Creutzfeldt-Jakob Disease, Down syndrome, etc.).
  2. Other neurodegenerative condition (amyotrophic lateral sclerosis, etc.).
  3. Seizure disorder.
  4. Other infectious, metabolic or systemic diseases affecting the central nervous system (syphilis, present hypothyroidism, present vitamin B12 or folate deficiency, other laboratory values etc.).
* Any major psychiatric diagnosis, including schizophrenia, bipolar disorder, and current major depressive disorder as per Diagnostic and Statistical Manual of Mental Disorders Fifth Edition
* Clinically significant, advanced or unstable disease that may interfere with outcome evaluations.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-05-19 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of CT1812 | Baseline, Day 1, Day 14, Day 28, Day 42, Day 56, Day 70, Day 98, Day 126, Day 154, Day 182, Day 210
  Incidence and Severity of Adverse Events

SECONDARY OUTCOMES:
Montreal Cognitive Assessment Scale (MoCA) | Baseline, 3 months, 6 months
  MOCA is a dementia screening assessment with a 0-30 range with lower scores meaning more impairment
Epworth Sleepiness Scale (ESS) | Baseline, 3 months, 6 months
  The ESS is an assessment of subjective sleepiness over the prior two weeks. The scale is on 4 point scale (0 = no chance of dozing; 1 = slight chance of dozing; 2 = moderate chance of dozing; 3 = high chance of dozing) An ESS score > 10 is considered consistent with excessive daytime sleepiness
Clinician Assessment of Fluctuation (CAF) | Baseline, 3 months, 6 months
  Assessment of cognitive fluctuations, with range of 1-16, with higher scores representing more severe fluctuations
ADCS-Clinical Global Impression of Change (CGIC) | Baseline, 3 months, 6 months
  The ADCS-CGIC is a 7-point scale similar to other global change scales, where a higher score indicates marked improvement
ADCS - Activities of Daily Living (ADCS-ADL) | Baseline, 3 months, 6 months
  Assessment of functional impairment in activities of daily living. The total score range is from 0-78 with lower scores indicating greater functional impairment.
Movement Disorder Society - United Parkinson's Disease Rating Scale Part III (MDS-UPDRS Part III) | Baseline, 3 months, 6 months
  This exam covers 18 motor signs associated with parkinsonism covering bradykinesia, rigidity, tremor, and gait with a range of scores from 0-136, with higher scores supporting more severe symptoms. A score of 6 or greater suggest the presence of parkinsonism
Cognitive Drug Research Battery (CDR) | Baseline, 3 months, 6 months
  Computerized battery that captures reaction time, cognitive reaction time, vigilance, and power of attention
Neuropsychiatric Inventory (NPI) | Baseline, 3 months, 6 months
  Assessment of common behaviors associated with dementia

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Caggiano, MD, Study Director — Cognition Therapeutics Inc.
Locations (34):
- United States (34):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - University of Arizona - Health Sciences Center, Tucson, Arizona
  - Stanford University, Palo Alto, California
  - Pacific Neuroscience Institute, Santa Monica, California
  - University of Colorado, Aurora, Colorado
  - CenExel Rocky Mountain Clinical Research, LLC, Englewood, Colorado
  - New England Institute for Neurology and Headache (NEINH), Stamford, Connecticut
  - JEM Research Institute, Atlantis, Florida
  - University of Miami Miller School of Medicine Comprehensive Center for Brain Health, Boca Raton, Florida
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Charter Research, Lady Lake, Florida
  - Renstar Medical Research, Ocala, Florida
  - Charter Research, Winter Park, Florida
  - Rush University Medical Center Section of Parkinson Disease and Movement Disorder, Chicago, Illinois
  - IU Health Neuroscience Center, Goodman Hall, Indianapolis, Indiana
  - Josephson Wallack Munshower Neurology, P.C, Indianapolis, Indiana
  - The University of Kansas Alzheimer's Disease Research Center, Fairway, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Headlands Research Eastern Massachusetts, LLC, Plymouth, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Columbia University, New York, New York
  - UNC Department of Neurology, Chapel Hill, North Carolina
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Summit Headlands, LLC, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - Clinical Trial Network, Houston, Texas
  - University of Virginia Adult Neurology, Charlottesville, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Evergreen Health Research, Kirkland, Washington
  - Universtiy of Washington Department of Neurology, Seattle, Washington

REFERENCES:
- [Derived] Galvin JE, Tolea MI, Scharre DW, Hamby ME, Iaci JF, Grundman M, Caggiano AO. Phase 2 study of zervimesine (CT1812) in participants with mild-to-moderate dementia with Lewy bodies (DLB). Alzheimers Dement. 2025 Dec;21(12):e71004. doi: 10.1002/alz.71004. PMID 41416579